CLINICAL TRIAL: NCT01365923
Title: Comparison of Dexmedetomidin and Remifentanil for the Effect on Airway Reflex and Hemodynamic Response During Emergence in Patients Undergoing Craniotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1-2011-0019
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2013-11

CONDITIONS: Open Craniotomy
MeSH Terms: interventions — Remifentanil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remifentanil group (Active Comparator): Remifentanil group : remifentanil effect site-TCI 2-4ng/ml
  Interventions: Drug: remifentanil
- Dexmedetimidine group (Active Comparator): Dexmedetomidine group: remifentanil effect site-TCI 2-4ng/ml + dexmedetomidine 0.5mcg/kg
  Interventions: Drug: dexmedetomidine with remifentanil

INTERVENTIONS:
Drug: remifentanil — remifentanil effect site-TCI 2-4ng/ml
  Arms: Remifentanil group
Drug: dexmedetomidine with remifentanil — remifentanil effect site-TCI 2-4ng/ml with dexmedetomidine 0.5mcg/kg
  Arms: Dexmedetimidine group

SUMMARY:
During recovery from general anesthesia the stimuli of endotracheal tube lead to the coughing, hypertension, tachycardia, which can cause a serious complication. Especially the postoperative course of patients emerging from general anesthesia after intracranial surgery is frequently complicated by the occurrence of hypertension and coughing event.

It has been demonstrated that opioid, intravenous or topical lidocaine administration can attenuate the coughing reflex. Administered the opioid before emergence, it is effective to prevent cough reflex but the recovery is delayed, it was difficult to predict emergence.

However, remifentanil is an opioid widely used because of rapid context-sensitive half-life, target-controled infusion method to adequately maintain the effect site concentration could help to predict the recovery time to the alert state from the general anesthesia. It is considered proper method of continuous infusion of remifentanil for reducing emergence cough.

Dexmedetomidine , a potent alpha adrenoceptor agonist which dose-dependently reduces arterial blood pressure and heart rate, decreases the hemodynamic and and catecholamine response to intubation and extubation. It is thus theologically appropriate for reducing airway and circulatory reflexes during emergence from anesthesia.

In this study, the investigators used bolus dexmedetomidine immediately before extubation, and compared the effects on coughing, hemodynamic response and recovery profile to a continuous infusion of remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* SA I~II, 2.aged between 20 and 70 year, 4.general anesthesia for craniectomy

Exclusion Criteria:

* signs of an anatomical or functional abnormality in upper airway
* URI or sore throat for recent 2 weeks
* Congestive heart failure, Sinus Bradycardia(<50 BPM), Uncontrolled hypertension
* Chronic obstructive lung disease, bronchial asthma

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
cough incidence | 1 minute after extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea